CLINICAL TRIAL: NCT06753864
Title: A Single-center, Open, Randomized, Single-dose, Cross-over Bioequivalence Study to Evaluate the Effects of the Test Formulation Abalparatide Injection and the Reference Formulation Abalparatide Injection (Tymlos®) in Healthy Adult Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Cao Yu, Director of the Phase I Clinical Research Center, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QLCG2128-01
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (T)-Reference (R） (Experimental): In this trial, 16 healthy subjects are planned to be enrolled in fasting. According to the randomization table, subjects will be randomly assigned to the Group A: Test (T)-Reference (R), The washout period (dosing interval) between doses will be at least 2 days. After fasting for at least 10 hours.
  Interventions: Drug: Test (T); Drug: Reference (R)
- Reference (R)-Test (T) (Experimental): In this trial, 16 healthy subjects are planned to be enrolled in fasting. According to the randomization table, subjects will be randomly assigned to the Group B: Reference (R)-Test (T), The washout period (dosing interval) between doses will be at least 2 days. After fasting for at least 10 hours.
  Interventions: Drug: Test (T); Drug: Reference (R)

INTERVENTIONS:
Drug: Test (T) — Abaloparatide injection, specification :3120 μg/1.56 ml(2000 μg/ml), drug information subject to actual supply, Qilu Pharmaceutical Co., LTD. The test preparations for the subjects are all from the same batch number.
Drug: Reference (R) — Abaloparatide injection (Tymlos®), specification :3120 μg/1.56 ml(2000 μg/ml), drug information is subject to actual supply, provided by Qilu Pharmaceutical Co., LTD. The reference preparations for the subjects were all from the same batch number.

SUMMARY:
To investigate the pharmacokinetics of the test preparation abalparatide injection and the reference preparation abalparatide injection (Tymlos®) in healthy adult subjects under fasting state, and to evaluate the bioequivalence of the two formulations under fasting state.

ELIGIBILITY:
Inclusion Criteria:

* 1. Before the test, voluntarily sign informed consent, fully understand the test content, process and possible adverse reactions, and complete the study according to the requirements of the test plan; 2. Female subjects have taken effective contraceptive measures within 14 days before the first dose (self-screening period for male subjects) and are willing to have no pregnancy, sperm donation or egg donation plan from signing informed to 6 months after the last dose, and voluntarily take effective contraceptive measures, specific contraceptive measures are shown in Appendix 2; 3. Male and female subjects aged 40 to 65 years (including boundary values); 4. Male subjects weigh no less than 50.0kg, female subjects weigh no less than 45.0kg, body mass index in the range of 19.0~28.0 kg/m2 (including the critical value).

Exclusion Criteria:

* 1. Have a history of serious diseases such as heart, liver, kidney, digestive tract, nervous system, endocrine system, respiratory system and mental disorders, which are considered unsuitable by the study doctor; 2. Clinically significant abnormalities judged by clinicians, including physical examination, vital signs examination, electrocardiogram or clinical laboratory examination; 3. Currently suffering from allergic diseases (urticaria, asthma, etc.), or allergies (such as allergies to two or more drugs, foods such as milk or pollen), or known allergies to components or analogues of the drug; 4. Patients with hyperparathyroidism, Paget's disease or history; 5. Past or present postural hypotension or dizziness in the morning; 6. Hyperuricemia (including previous history of gout), hypercalcemia or active urinary calculus; 7. Serum calcium higher than the upper limit of normal, or creatinine clearance <80mL/min(calculation formula: male Ccr(mL/min)= [(140- age)× body weight (kg)]/[0.818× serum creatinine (μmol/L)]; Ccr female =Ccr male ×0.85); 8. Patients who have previously received extra-skeletal beam or implanted radiation therapy; 9. Female subjects who are pregnant, breastfeeding or have positive pregnancy test results; 10. Hepatitis B surface antigen, hepatitis C antibodies, HIV antibodies or syphilis antibodies, any one or more of which are positive 11. Have a history of drug abuse within 5 years, or have used drugs within 3 months before screening, or urine drug screening is positive; 12. Those who consumed an average of more than 14 units of alcohol per week (1 unit =360mL beer or 45mL liquor with 40% alcohol or 150mL wine) in the 3 months prior to screening, or who could not stop alcohol intake from 24h before first dosing to the completion of all blood samples collected, or who tested positive for alcohol breath tests; 13. Those who smoked more than 5 cigarettes per day in the 3 months before screening or stopped using tobacco products during the period of refusal to stay; 14. Had a history of surgery within 3 months prior to screening, or planned to have surgery during the study period; 15. Those who donated blood or lost a lot of blood within 3 months before the first administration (>400mL, except for female physiologic blood loss), or donated platelets ≥2 therapeutic amounts (1 therapeutic amount =12U platelets) within 1 month; 16. Participants in any drug clinical trial and administration within 3 months before the first dose; 17. Those who have received any prescription drugs (including vaccines) within 14 days prior to the first dose; 18. Those who have received any over-the-counter medicines (including birth control pills), Chinese herbs or health products (including vitamins) within 7 days before the first dose; 19. ngested any food rich in xanthines (such as coffee, tea, chocolate, cocoa, milk tea, etc.), grapefruit (grapefruit), pomelo, pomegranate, lime, star fruit and its products, or had intense exercise, or other factors affecting drug absorption, distribution, metabolism, excretion, etc.; 20. Patients with difficulty in venous blood collection or a history of fainting needles and fainting blood, or skin scars, wounds or tattoos at the injection site, which affect the absorption or observer of injection drugs; 21. Subjects deemed unsuitable for participation by other investigators.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-02 (Estimated); Primary Completion 2025-01-09 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 4 hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t） | 4 hours
  Area under the drug concentration-time curve from time 0 to the 4h accurately measurable concentration at sample collection time
Area under the plasma concentration versus time curve (AUC0-∞) | 4 hours
  Area Under the Plasma Drug Concentration-Time Curve from Time 0 to Infinite Time

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No